CLINICAL TRIAL: NCT00453960
Title: Effect of Genistein on Endometrial Hyperplasia
Brief Title: Genistein and Endometrial Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: University of Messina, University of Messina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Roberta Granese, MD, PhD
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2008-12-19 (Estimated); Status verified 2008-12

CONDITIONS: Endometrial Hyperplasia
Keywords: Endometrial hyperplasia; Genistein; Isoflavones; dysfunctional uterine bleeding
MeSH Terms: conditions — Endometrial Hyperplasia; Metrorrhagia | interventions — Norethindrone Acetate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Genistein (Experimental): Genistein 54 mg/day
  Interventions: Dietary Supplement: Genivis
- Norethisterone Acetate (Active Comparator): Norethisterone Acetate 10mg/day
  Interventions: Drug: Norethisterone Acetate
- Placebo (Placebo Comparator): Placebo tablets, daily
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Genivis — 54 mg/day daily for 6 months
  Other Names: Fosteum
  Arms: Genistein
Drug: Norethisterone Acetate — tablets 10mg/day from day 16 to 25 of menstruation
  Arms: Norethisterone Acetate
Other: placebo — tablets daily for 6 months
  Arms: Placebo

SUMMARY:
The aim of this study is to verify the anti-estrogenic activity of Genistein, on the "non atypical endometrial hyperplasia", in premenopausal women.

DETAILED DESCRIPTION:
Although isoflavones alone (example: Genistein) have weak estrogenic effects on endometrial stromal and glandular cells, it was demonstrated, in several research efforts, that in the presence of E2 they act as antiestrogens.

Considered that endometrial hyperplasia is due to strong and extended estrogenic stimulation, not offset by a proportionate amount of progesterone, we suppose that genistein could be therapeutic in these cases inducing a decrease of the hyperplasia and a change from the proliferative to a secretory phase of the endometrium.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women
* Age > = 44 years
* Dysfunctional uterine bleeding
* No treatment with other hormonal drugs (estrogen, progesterone)
* No local or general pathology negatively influenced by administration of genistein or progesterone
* No intrauterine pathologies (polyps, myomas)
* A "non atypical endometrial hyperplasia", confirmed by hysteroscopy with biopsy and histological examination

Exclusion Criteria:

* All the other conditions

Ages: 44 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2007-01; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Recovery from endometrial hyperplasia | 3-6 months

SECONDARY OUTCOMES:
Differential expression of ER-a and ER-b in endometrial specimens | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rosario D'Anna, prof., Study Director — menopause centre
Locations (1):
- Menopause Centre, Department of Gynecology and Obstetrics, Policlinico Universitario "G.Martino", Messina, Italy

REFERENCES:
- [Result] Kayisli UA, Aksu CA, Berkkanoglu M, Arici A. Estrogenicity of isoflavones on human endometrial stromal and glandular cells. J Clin Endocrinol Metab. 2002 Dec;87(12):5539-44. doi: 10.1210/jc.2002-020716. PMID 12466350